CLINICAL TRIAL: NCT03979703
Title: Effectiveness of Yoga in Patients With Fibrosing Interstitial Lung Diseases - a Feasibilty and Pilot Study
Brief Title: Yoga in Patients With Fibrosing Interstitial Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Lungenfibrose e.V. (Unknown)
Responsible Party: Principal Investigator, Michael Kreuter, Principal Investigator, Clinical Professor, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Yoga-Study
Record Dates: First submitted 2019-05-14; First posted 2019-06-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Fibrosing Interstitial Lung Diseases; Idiopathic Pulmonary Fibrosis
Keywords: fibrosing interstitial lung disease; Idiopathic Pulmonary Fibrosis; Yoga
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention will be a 12 week yoga class
  Interventions: Other: 12 week yoga class
- Control group (No Intervention): Control group will not participate in the 12 week yoga class but will participate in Surveys, 6 minute walking test, lung function test, and biomarker analysis. Furthermore, they will be offered a yoga class after the study.

INTERVENTIONS:
Other: 12 week yoga class — Intervention is a 12 week yoga class with classes twice a week. Each yoga class will last about 1 hour. Furthermore, focus group interviews will be conducted after the first and last yoga class.
  Arms: Intervention group

SUMMARY:
Fibrosing interstitial lung diseases are characterized by loss of lung function, which leads to a decrease in quality of life and physical capacity. Several studies have shown an increase in quality of life and physical capacity after increasing physical activity in patients. There is evicence that yoga has a positive influence in patients with chronic obstructive pulmonary diseases, but so far, studies examining the effect of yoga in patients with fibrosing interstitial lung diseases are missing.

Study aims are to determine the feasibilty of this study, and to determine the effects of yoga to patients' quality of life and physical capacity.

Twenty patients with a fibrosing interstitial lung disease will be recruited and randomly assigned to the intervention or control group. Several questionnaires regarding quality of life will be conducted. Furthermore, the 6 minutes walking test, a lung function test and a biomarker analysis will be conducted at baseline and follow-up. The intervention group will participate in a 12 week yoga class, whereas the controll group will not participate. Yoga classes will be offered to the control group after the study.

In addition, focus group interviews will be conducted at baseline and follow-up with the intervention group.

DETAILED DESCRIPTION:
Patients with a fibrosing interstitial lung disease will be recruited. In total 20 patients will be recruited, 10 for the intervention group and 10 for the control group.

The Intervention group will participate in a 12 week yoga class with classes twice a week for about 1 hour. The control group will not participate in a yoga class.

At baseline all patients will conduct a 6 minutes walking test, a lung function test, several surveys to measure health related quaility of life (King's Brief Interstitial Lung Disease Questionnaire (K-BILD), Hospital Anxiety and Depression Scale (HADS), Interstitial Lung Disease Anxiety questionnaire), and some blood will be drawn for biomarker analysis.

Furthermore, participants in the Intervention group will participate in two focus group interviews, one at baseline and the second one at 12 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand study and study procedure
* diagnosis of fibrosing interstitial lung disease
* Age: > 18 years
* Ability to consent

Exclusion Criteria:

* Forced Vital Capacity < 50%
* Oxygen therapy
* diagnosis of pulmonary hypertension
* participant does not understand the study
* pulmonary infection within the last 4 weeks
* acute exacerbation within the last 4 weeks
* other respiratory decline within the last 4 weeks
* co-morbidities which make yoga training impossible

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of life at 12 weeks: King's Brief Interstitial Lung Disease Questionnaire (K-BILD) | baseline and 12 week follow-up
  Quality of life will be measured with King's Brief Interstitial Lung Disease Questionnaire (K-BILD). It is a 15-item validated questionnaire assessing health status in patients with an interstitial lung disease. Questions are related to three domains: breathlessness and activities, psychological aspects, and chest symptoms. Each question has 7 possible answers. The questionnaire has a scale from 0 - 100, in which 100 means highest quality of life.
Change in physical capacity | baseline and 12 week follow-up
  Physical capacity will be measured by the 6 miuntes walking test
Feasibility of a yoga class in patients with fibrosing interstitial lung diseases: focus group interview | 12 week follow-up
  Evaluation of the study by a focus group interview
Change from baseline quality of life at 12 weeks: Hospital Anxiety and Depression Scale (HADS) | baseline and 12 week follow-up
  Quality of life will be measured with the Hospital Anxiety and Depression Scale (HADS). It is a 14-item questionnaire, 7 items are related to depression and 7 items are related to anxiety. Each question has 4 different answer options, each scored from 0-3. Scores are summed up for each field (depression or anxiety) with 0 points as lowest possibility and 21 scores as highest (0-7 = normal, 8-10 = borderline abnormal, and 11-21 = abnormal).
Change from baseline quality of life at 12 weeks: Interstitial Lung Disease Anxiety-questionnaire | baseline and 12 week follow-up
  Quality of life will be measured with Interstitial Lung Disease Anxiety-questionnaire. This is a 37-item questionnaire with 5 answer possibilities for each question (never, rare, sometimes, often, always). Total scores are a sum of all questions. Lowest score = 0, highest score = 136. The higher the score the better is the patients' quality of life.
Expectations of study by participants | baseline
  Evaluation of the study by a focus group interview

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kreuter, Prof., Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik-Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No